CLINICAL TRIAL: NCT07348822
Title: 8-Year Outcomes After Sleeve Gastrectomy: Anthropometric, Biochemical, and Nutritional Evaluation
Brief Title: 8-Year Outcomes After Sleeve Gastrectomy
Status: Active, not recruiting | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Seher Şen, Assist. Prof. Dr., Medipol University
Other Study IDs: MUDU-SBE-SS-02
Record Dates: First submitted 2025-12-18; First posted 2026-01-16 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Sleeve Gastrectomy; Obesity & Overweight
Keywords: long-term follow-up; sleeve gastrectomy; obesity; metabolic outcomes; nutritional status; anthropometric measurements
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sleeve Gastrectomy Long-Term Follow-up Cohort: This cohort includes adults who underwent sleeve gastrectomy between 2016 and 2017 and were re-evaluated approximately 8 years after surgery. Participants are followed observationally, with anthropometric measurements, biochemical parameters, and nutritional status assessed preoperatively, at postoperative 6 months, and at long-term (8-year) follow-up. No intervention is assigned as part of the study protocol; all surgical procedures were performed as part of routine clinical care.

SUMMARY:
Obesity is a major global public health concern, and bariatric surgery is recognized as the most effective treatment for achieving sustained weight loss and improving obesity-related comorbidities. Sleeve gastrectomy (SG) is one of the most commonly performed bariatric procedures; however, long-term outcomes vary considerably among individuals. While some patients maintain satisfactory weight loss, others experience suboptimal weight loss or weight regain several years after surgery. Evidence suggests that long-term weight trajectories after SG may be influenced by metabolic changes, dietary habits, and lifestyle factors, highlighting the need for extended follow-up studies.

This observational cohort study aims to evaluate the long-term outcomes of individuals who underwent sleeve gastrectomy approximately 8 years ago. Anthropometric measurements, biochemical parameters, and nutritional status will be reassessed at an 8-year follow-up visit and compared with data obtained during the preoperative period and at postoperative 6 months. By examining within-subject changes over time, this study seeks to provide insight into the long-term sustainability of weight loss after sleeve gastrectomy and to identify metabolic and nutritional factors associated with long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* Patients who underwent sleeve gastrectomy approximately 8 years prior to study enrollment
* Patients with available postoperative follow-up data at 6 months, including anthropometric measurements, biochemical parameters, and nutritional status assessments
* Patients willing to participate in long-term follow-up and attend in-person evaluations

Exclusion Criteria:

* Pregnancy or lactation
* Presence of acute illness or active infection at the time of evaluation
* Presence of acute illness, infection, or comorbid conditions that may limit study safety or validity, including malignancy, type 1 diabetes mellitus, renal or hepatic failure, recent stroke or myocardial infarction, nephrolithiasis, drug or alcohol abuse, eating disorders, severe depression or other major psychiatric disorders, inflammatory bowel disease, cardiac arrhythmias or heart failure, respiratory failure, or chronic systemic corticosteroid therapy.
* Professional athletes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adults aged 18-65 years who underwent sleeve gastrectomy approximately eight years prior to enrollment and completed standard postoperative follow-up. Participants had available preoperative and 6-month postoperative anthropometric, biochemical, and nutritional data and were re-evaluated at 8 years after surgery to assess long-term outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2026-01-10 (Actual); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Change in Fat Mass | Preoperative, postoperative 6 months, and postoperative 8 years
  Changes in fat mass measured using multi-frequency bioelectrical impedance analysis (BIA).
Change in Body Weight | Preoperative, postoperative 6 months, and postoperative 8 years
  Body weight measured using a calibrated digital scale with participants wearing light clothing and no shoes.
Change in Body Mass Index (BMI) | Preoperative, postoperative 6 months, and postoperative 8 years
  BMI calculated as weight in kilograms divided by height in meters squared (kg/m²), measured using a wall-mounted stadiometer.
Change in Waist Circumference | Preoperative, postoperative 6 months, and postoperative 8 years
  Waist circumference measured in centimeters at the midpoint between the subcostal margin and the iliac crest with participants standing upright.
Change in Hip Circumference | Preoperative, postoperative 6 months, and postoperative 8 years
  Hip circumference measured in centimeters at the level of maximum gluteal protrusion.
Percent Total Weight Loss (TWL%) | Postoperative 6 months and postoperative 8 years
  Calculated as [(preoperative weight - postoperative weight) / preoperative weight] × 100.
Percent Excess Weight Loss (EWL%) | Postoperative 6 months and postoperative 8 years
  Calculated as [(preoperative weight - postoperative weight) / (preoperative weight - ideal body weight)] × 100, where ideal body weight corresponds to a BMI of 25 kg/m².
Change in Body Fat Percentage | Preoperative baseline, postoperative 6 months, and postoperative 8 years
  Changes in body fat percentage measured using multi-frequency bioelectrical impedance analysis (BIA).
Change in Skeletal Muscle Mass | Preoperative baseline, postoperative 6 months, and postoperative 8 years
  Changes in skeletal muscle mass measured using multi-frequency bioelectrical impedance analysis (BIA).

SECONDARY OUTCOMES:
Change in Fasting Plasma Glucose | Preoperative, postoperative 6 months, and postoperative 8 years
  Fasting plasma glucose measured after at least 8 hours of fasting using venous blood samples.
Change in Fasting Insulin Levels | Preoperative, postoperative 6 months, and postoperative 8 years
  Fasting insulin levels measured from venous blood samples obtained after at least 8 hours of fasting.
Change in Glycated Hemoglobin (HbA1c) | Preoperative, postoperative 6 months, and postoperative 8 years
  HbA1c levels measured to assess long-term glycemic control.
Change in Lipid Profile Parameters | Preoperative, postoperative 6 months, and postoperative 8 years
  Serum lipid parameters including total cholesterol, LDL cholesterol, HDL cholesterol, and triglycerides measured after an overnight fast.
Change in Liver Enzyme Levels | Preoperative, postoperative 6 months, and postoperative 8 years
  Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels measured from fasting blood samples.
Change in Renal and Metabolic Biomarkers | Preoperative, postoperative 6 months, and postoperative 8 years
  Serum urea and uric acid levels measured to assess renal and metabolic function.
Change in Serum Albumin | Preoperative, postoperative 6 months, and postoperative 8 years
  Changes in serum albumin levels measured from venous blood samples.
Change in Micronutrient Levels | Preoperative, postoperative 6 months, and postoperative 8 years
  Serum levels of vitamin B12, folic acid, magnesium, total calcium, sodium, and potassium measured to assess micronutrient status.
Change in Physical Activity Level | Preoperative, postoperative 6 months, and postoperative 8 years
  Physical activity levels assessed using the International Physical Activity Questionnaire (IPAQ).
Change in Fat-Free Mass | Preoperative baseline, postoperative 6 months, and postoperative 8 years
  Changes in fat-free mass measured using multi-frequency bioelectrical impedance analysis (BIA).
Change in Total Protein | Preoperative baseline, postoperative 6 months, and postoperative 8 years
  Changes in total serum protein levels measured from venous blood samples.
Change in Hemoglobin | Preoperative baseline, postoperative 6 months, and postoperative 8 years
  Changes in hemoglobin levels measured from venous blood samples.
Change in Hematocrit | Preoperative baseline, postoperative 6 months, and postoperative 8 years
  Changes in hematocrit levels measured from venous blood samples.
Change in Serum Ferritin | Preoperative baseline, postoperative 6 months, and postoperative 8 years
  Changes in serum ferritin levels measured from venous blood samples.
Change in Serum Iron | Preoperative baseline, postoperative 6 months, and postoperative 8 years
  Changes in serum iron levels measured from venous blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Seher Şen, Study Director — Mudanya University
Locations (1):
- Mudanya Univesity, Bursa, Mudanya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the need to protect patient privacy and confidentiality. T